CLINICAL TRIAL: NCT02619019
Title: Intrathecal Dexamethasone in Patients Undergoing Transuretheral Prostatectomy.
Brief Title: Effect of Spinal Dexamethasone During Transuretheral Prostatectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Seham Mohamed Moeen Ibrahim, lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SM112015
Record Dates: First submitted 2015-11-27; First posted 2015-12-02 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Postspinal Shivering
MeSH Terms: interventions — Dexamethasone; Meperidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dexamethasone group (Active Comparator): Patients will receive 8 mg of hyperbaric bupivacaine 0.5%, plus 8 mg of dexamethasone intrathecally
  Interventions: Drug: Dexamethasone
- Pethidine group (Active Comparator): Patients will receive 8 mg of hyperbaric bupivacaine 0.5%, plus 0.2 mg/kg of pethidine intrathecally
  Interventions: Drug: Pethidine
- Control group (Placebo Comparator): Patients will receive 8 mg of hyperbaric bupivacaine 0.5%, plus 2 ml normal saline intrathecally
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexamethasone — Patients will receive 8 mg of hyperbaric bupivacaine 0.5%, plus 8 mg of dexamethasone intrathecally
  Arms: Dexamethasone group
Drug: Pethidine — Patients will receive 8 mg of hyperbaric bupivacaine 0.5%, plus 0.2 mg/kg of pethidine intrathecally
  Other Names: Mepredine
  Arms: Pethidine group
Drug: Normal saline — Patients will receive 8 mg of hyperbaric bupivacaine 0.5%, plus 2 ml normal saline intrathecally
  Arms: Control group

SUMMARY:
Dexamethasone, a high-potency, long-acting glucocorticoid, when added to bupivacaine, it extended the duration of analgesia. We aim to study the effectiveness of spinal dexamethasone in Transuretheral prostatectomy.

DETAILED DESCRIPTION:
Spinal anesthesia for endoscopic urology surgery like transurethral resection of the prostate is a well-established technique. Opioids are extensively used as an adjunct to local anesthetics in neuraxial blockade to enhance the duration of postoperative analgesia. However, worrisome adverse effects like pruritus, urinary retention, postoperative vomiting and respiratory depression limit its use. The aim of this study was to investigate the effectiveness of Intrathecal dexamethasone as adjunct to local anesthetics.

ELIGIBILITY:
Inclusion Criteria:

* Age: 50-75 yr ASA class I,II, and III undergoing Transuretheral prostatectomy under spinal anesthesia

Exclusion Criteria:

* Contraindications to spinal anesthesia, Allergy to the study medication, Thyroid disease, Parkinson's disease Patients receiving vasodilators or medications likely to alter thermoregulation.

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Shivering | 150 min after spinal anesthesia
  by shivering score

SECONDARY OUTCOMES:
Mean arterial blood pressure | 150 min after spinal anesthesia
  immediately before the block and then every 15 min after the block
Heart rate | 150 min after spinal anesthesia
  immediately before the block and then every 15 min after the block
Core temperature | 150 min after spinal anesthesia
  immediately before the block and then every 15 min after the block

CONTACTS AND LOCATIONS:
Overall Officials: Seham M Moeen, MD, Principal Investigator — Assiut Univerisity
Locations (1):
- Seham Mohamed Moeen Ibrahim, Asyut, Asyut Governorate, Egypt